CLINICAL TRIAL: NCT02287623
Title: Subcostal TAP Block With Liposomal Bupivacaine vs Bupivacaine in Donor Nephrectomy Patients: A Prospective Randomized Study
Brief Title: Subcostal TAP Block With Liposomal Bupivacaine Versus Bupivacaine in Donor Nephrectomy Patients: A Prospective Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1301M27261
Record Dates: First submitted 2014-10-30; First posted 2014-11-11 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- liposomal bupivacaine TAP (Experimental): Patients will receive a TAP block with liposomal bupivacaine
  Interventions: Drug: liposomal bupivacaine
- bupivacaine TAP (Active Comparator): Patients will receive a TAP block with bupivacaine
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: liposomal bupivacaine — patients will receive a tap with liposomal bupivacaine
  Arms: liposomal bupivacaine TAP
Drug: bupivacaine — patients will receive a tap with bupivacaine
  Arms: bupivacaine TAP

SUMMARY:
The primary objective of this study is whether one local anesthetic, liposomal bupivacaine, provides improved pain control and decreased opioid use compared to bupivacaine when injected during a transversus abdominis plane block for donor nephrectomy patients.

DETAILED DESCRIPTION:
The primary objective of this study is whether one local anesthetic, liposomal bupivacaine, provides improved pain control and decreased opioid use compared to bupivacaine when injected during a transversus abdominis plane block for donor nephrectomy patients.

Background and treatment procedure: Liposomal bupivacaine is a multi vesicular formulation of bupivacaine that has been shown to provide up to 72 hours of analgesia compared to bupivacaine which provides up to 24 hours of analgesia post injection. These two medications have been compared using a infiltration or injection at the site of incision but have yet to be compared when used during a TAP block. A TAP block is an injection of local anesthetic under the covering of the transversus abdominis muscle layer. This layer is found using an ultrasound which is a beam of high frequency sound that allows one to visualize images in the body. Then using this ultrasound we can see our needle as it pierces the covering of the transversus abdominis muscle layer and watch as the local anesthetic is injected into this plane. This is done on both sides of the abdomen to provide analgesia to the skin, muscle, and fascial layers of the abdomen.

Population: Adult patients who are undergoing a donor nephrectomy Rationale: It will be useful to determine if one formulation or the other provides better and longer lasting pain control for patients undergoing abdominal procedures.

ELIGIBILITY:
Inclusion Criteria:

* presenting for donor nephrectomy

Exclusion Criteria:

* non english speaking
* chronic pain condition
* taking chronic opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine TAP: Patients will receive a TAP block with liposomal bupivacaine
  liposomal bupivacaine: patients will receive a tap with liposomal bupivacaine in the preoperative area before the kidney donation. This occurred under ultrasound guidance with the patient sedated. the patient received 30 mL total per tap. Each TAP consisted of 10 mL of liposomal bupivacaine and 20 mL of normal saline.
- Bupivacaine TAP: Patients will receive a TAP block with bupivacaine bupivacaine: patients will receive a tap with bupivacaine in the preoperative area before the kidney donation. This occurred under ultrasound guidance with the patient sedated. the patient received 30 mL total per tap. Each TAP consisted of 30 mL of 0.25% bupivacaine with 1:200,000 epinephrine.
Period: Overall Study
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: we analyzed patients age, weight and gender.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 57
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59
weight [Mean (Standard Deviation); unit: kilograms] | 78.7 (12.3) | 75.5 (15.5) | 77.1 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale
Description: This was a measure of patient's reported pain on a 0-10 verbal numerical rating scale. 10 being worst pain. The maximal value for the time period 48-72 hours was chosen as the maximal pain during that time period.
Time Frame: 48-72 hours after injection
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Number analyzed (Participants) | 30 | 29
scores on a scale | 5 [3 to 7] | 3 [2 to 5]

2. Secondary Outcome: Post Operative Opioid Use
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: micrograms of fentanyl equivalents
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Number analyzed (Participants) | 30 | 29
micrograms of fentanyl equivalents | 70 [30 to 170] | 170 [65 to 250]

3. Secondary Outcome: Number of Patients With Post Operative Nausea/Vomiting
Time Frame: 0-72 hours
Measure: Number; unit: participants
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Number analyzed (Participants) | 30 | 29
participants | 7 | 15

4. Secondary Outcome: Post Operative Length of Stay
Time Frame: up to 30 days after surgery
Measure: Median (Inter-Quartile Range); unit: HOURS
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Number analyzed (Participants) | 30 | 29
HOURS | 67.7 [55.4 to 77.8] | 78.1 [62.8 to 82.3]

5. Secondary Outcome: Postoperative Opioid Use
Description: Use of opioids during 24-48 hours after surgery
Time Frame: 24-48 hours
Measure: Median (Inter-Quartile Range); unit: Micrograms of fentanyl equivalents
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Number analyzed (Participants) | 30 | 29
Micrograms of fentanyl equivalents | 190 [100 to 335] | 240 [125 to 375]

6. Secondary Outcome: Post Operative Opioid Use
Description: Post operative opioid use from 0-24 hours after surgery.
Time Frame: 0-24 hours
Measure: Median (Inter-Quartile Range); unit: micrograms of fentanyl equivalents
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Number analyzed (Participants) | 30 | 29
micrograms of fentanyl equivalents | 160 [107.5 to 322.5] | 230 [100 to 315]

ADVERSE EVENTS:
Arm/Group | Liposomal Bupivacaine TAP | Bupivacaine TAP
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes